CLINICAL TRIAL: NCT04986020
Title: Identifying New Biomarkers of Parkinson's From Routine Brain Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Stephen Mullin, Clinical Lecturer in Neurology, University of Plymouth
Other Study IDs: 2557; IRAS 280243 (Other: Health Research Authority)
Record Dates: First submitted 2021-07-21; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson disease: Participants with a clinical diagnosis of Parkinson's disease
  Interventions: Diagnostic Test: MRI
- Control: Controls
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Identification of novel biomarkers from MRI

SUMMARY:
The study will use routine computer tomography (CT), magnetic resonance spectroscopy (MRI) and nuclear medicine (NM) brain imaging data to produce new diagnostic tests for the onset of Parkinson's disease. This will enable hopefully earlier diagnosis than is currently possible. This will entail the analysis of anonymised CT/MRI/NM brain images collected prior to the point when these subjects were diagnosed with PD.

DETAILED DESCRIPTION:
We intend to use historical CT/MRI/nuclear medicine brain scans to identify novel imaging biomarkers of prodromal Parkinson's disease. The primary data source for the study will be MRI and CT brain scans, whilst nuclear medicine imaging brain imaging (DAT scans) will be used to validate models produced and provide a functional outcome measure of brain dopamine uptake. We shall utilise a an artificial intelligence approach to compare scans of PD cases with matched controls in order to identify these imaging biomarkers.

A list of participants with a diagnosis will be compiled. This list, together with relevant clinical data, will be linked with historical CT/MRI/nuclear medicine scans carried out over the preceding years. A control group of matched non-PD scans will also be compiled.

The dataset will be anonymised and a bespoke ML pipeline will be used to identify imaging featureswhich may be indicative of prodromal PD. This initial stage will be carried out at University Hospital Plymouth NHS Trust (UHPNT), the Royal Cornwall Hospital NHS Trust (RCHNT) and Cornwall Partnership NHS Trust (CPNT). If successful, findings will be validated in a larger sample of scans compiled from hospitals regionally and nationally.

ELIGIBILITY:
Inclusion Criteria:

- A clinical diagnosis of Parkinson's

Exclusion Criteria:

- No clinical diagnosis of Parkinson's

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants drawn from the catchment areas of participating healthcare organisations
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The presence of novel putative biomarkers of future PD development as defined by a deep-learning method | 3 years

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT04986020/Prot_000.pdf